CLINICAL TRIAL: NCT02122393
Title: A Randomised, Controlled Evaluation of Sertraline, Cognitive Behaviour Therapy & Combined Therapy for Postnatal Depression
Brief Title: A Randomised Trial of Sertraline, Cognitive Behaviour Therapy & Combined Therapy for Postnatal Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jeannette Milgrom, Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2001/01263
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sertraline (Active Comparator)
  Interventions: Drug: Sertraline
- Cognitive Behavioural Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Combined Therapy (Active Comparator)
  Interventions: Drug: Sertraline; Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Drug: Sertraline
  Arms: Combined Therapy; Sertraline
Behavioral: Cognitive Behavioural Therapy
  Arms: Cognitive Behavioural Therapy; Combined Therapy

SUMMARY:
Th purpose of this study is to determine whether dual psychological and pharmacological treatment is superior to either mono-therapy alone in the treatment of postnatal depression.

ELIGIBILITY:
Inclusion Criteria:

* Women with an infant > 2 months and < 8 months of age
* Infant born after a full-term pregnancy
* Infant born with no congenital abnormalities
* Diagnosis of depression with postnatal onset according to the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV).

Exclusion Criteria:

* positive serum pregnancy test;
* concurrent psychiatric disorder (excepting co-morbid anxiety);
* recent history of antidepressant usage (within the last month);
* history of major allergy or drug allergy;
* history of substance abuse;
* prior non-response to sertraline, or prior non-response to adequate trials of two selective serotonin reuptake inhibitors (SSRIs);
* predisposition to headache, migraine or nausea;
* tobacco habit in excess of 10 cigarettes per day;
* caffeine consumption in excess of 6 cups of coffee/tea or cola-flavoured drinks per day;
* ongoing dental work;
* extreme levels of depression (psychotic);
* suicidal intent;
* participation in any medical trial within the previous three months;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2002-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 24 weeks

SECONDARY OUTCOMES:
Beck Anxiety Inventory | 24 weeks
Parenting Stress Index | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Milgrom, PhD, Principal Investigator — University of Melbourne; Alan W Gemmill, PhD, Study Director — Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia